## Title:

Using narrow-band imaging (NBI) technique to detect post-radiotherapy mucosal residual nasopharyngeal carcinoma (NPC)

## **Principle Investigator**

Dr. Wong Kai Chuen,

## Statistical Analysis plan

- 1. Post-RT NP NBI vessel pattern were analyzed
- 2. Vessel pattern will be divided into NBI suspicious group and NBI non suspicious group
- 3. 2x2 table of suspicious/ non-suspicious group vs no residual disease / have residual disease will be obtained
- 4. Chi-square test will be performed, p-value will be contained
- 5. Sensitivity, specificity, positive predicted valve, negative predicted value of using NBI to detect mucosal residual NPC will be calculated